CLINICAL TRIAL: NCT04071249
Title: Validation of the Combined Symptom and Medication Score (CSMS) in Patients Suffering From Allergic Rhinoconjunctivitis Induced by Tree Pollen, Grass Pollen or House Dust Mites Who Are Treated Exclusively With Symptomatic Medication
Brief Title: Validation of a Combined Symptom and Medication Score in Patients Suffering From Allergic Rhinoconjunctivitis
Status: Completed | Type: Observational
Sponsor: ClinNovis GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: Control Validation CSMS 2019
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Rhinoconjunctivitis, Allergic
Keywords: Combined Symptom and Medication Score (CSMS); Validation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Control: Patients who use symptomatic medication as therapy for their allergic rhinoconjuntivitis as recommended by their physician

SUMMARY:
This study is a mere data collection without predefined intervention. Patients aged 12 years or older who suffer from allergic rhinitis induced by house dust mites, tree pollen or grass pollen and who are treated exclusively with anti-allergic medication may take part. The treatment follows the normal medical practice in accordance with national medical guidelines. During the study, data are collected during 3 visits with regard to allergic complaints of a patient and intake of anti-allergic medication. The first visit takes place before allergen exposure, the second visit at the peak of allergen exposure and the third visit after allergen exposure. The allergen exposure is defined as the enhanced exposure to house dust mites during the heating period or the respective pollen season. During the visits, the patients will be asked to complete questionnaires with regard to their quality of life and rhinitis control. Furthermore during allergen exposure, the patients document their allergic complaints and intake of anti-allergic medication in a diary. The diary entries are used to generate the Combined Symptom and Medication Score (CSMS) which will be validated in the course of this study. The validation will be performed by comparing the CSMS with the scores from the already validated questionnaires.

DETAILED DESCRIPTION:
This study is a prospective, mulit-center data collection without predefined intervention. Patients aged 12 years or older who suffer from allergic rhinoconjunctivitis induced by house dust mites, tree pollen or grass pollen and who are treated exclusively with symptomatic medication may take part. The treatment follows the normal medical practice in accordance with national medical guidelines. During the study, data are collected during 3 visits with regard to allergic symptoms of a patient and intake of symptomatic medication. The first visit takes place before allergen exposure, the second visit at the peak of allergen exposure and the third visit after allergen exposure. The allergen exposure ist defined as the enhanced exposure to house dust mites during the heating period or the respective pollen season. During the visits, the patients will be asked to complete questionnaires [the rhinitis quality of life questionnaire (RQLQ, Visit 1, 2 and 3) and the rhinitis control assessment test (RCAT, visit 2)]. Furthermore during allergen exposure, the patients document allergic symptoms and intake of symptomatic medication in a diary. These diary entries are used to generate the Combined Symptom and Medication Score (CSMS) which will be validated in the course of this study. The validation will be performed by comparing the CSMS with the scores from the already validated RQLQ and RCAT.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 12 years or older who suffer from allergic rhinoconjunctivitis induced by house dust mites, tree pollen or grass pollen and who are treated exclusively with symptomatic medication

Exclusion Criteria:

* Allergen-specific immunotherapy

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 12 years or older who suffer from allergic rhinoconjunctivitis induced by house dust mites, tree pollen or grass pollen and who are treated exclusively with symptomatic medication
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
Combined Symptom and Medication Score (CSMS) | 30 to 60 days during allergen exposure
  The CSMS describes the severity of nasal and conjunctival symptoms of allergic rhinoconjunctivitis as well as the intake of symptomatic medication.
  Four nasal and two conjunctival symptoms (itchy nose, sneezing, runny nose, blocked nose, itchy/red eyes, watery eyes) are evaluated using a score from 0 to 3 (0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms, 3 = severe symptoms).
  The stepwise use of medication will be assessed as follows:
  1. = Oral and/or topical (eyes or nose) nonsedative H1 antihistamines (H1A)
  2. = Intranasal corticosteroids (INS) with/without H1A
  3. = Oral corticosteroids with/without INS, with/without H1A
  The combination of symptom and medication score based on an equal weight generates the daily CSMS with a range from 0 to 6.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Moesges, Prof. Dr., Study Chair — ClinNovis GmbH, Genter Str. 7, 50672 Cologne, Germany
Locations (7):
- Germany (7):
  - Otorhinolaryngology practice, Aachen
  - Otorhinolaryngology practice, Bad Schönborn
  - Practice for lung and bronchial medicine, Bonn
  - Otorhinolaryngology practice, Dresden
  - Otorhinolaryngology practice, Duisburg
  - Otorhinolaryngology practice, Füssen
  - Otorhinolaryngology practice, Schorndorf

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pfaar O, Demoly P, Gerth van Wijk R, Bonini S, Bousquet J, Canonica GW, Durham SR, Jacobsen L, Malling HJ, Mosges R, Papadopoulos NG, Rak S, Rodriguez del Rio P, Valovirta E, Wahn U, Calderon MA; European Academy of Allergy and Clinical Immunology. Recommendations for the standardization of clinical outcomes used in allergen immunotherapy trials for allergic rhinoconjunctivitis: an EAACI Position Paper. Allergy. 2014 Jul;69(7):854-67. doi: 10.1111/all.12383. Epub 2014 Apr 25. PMID 24761804